CLINICAL TRIAL: NCT05785260
Title: Promoting and Supporting Mental and Physical Well-being: the Role of Smart Health in the Prevention of Cerebrocardiovascular Disease
Brief Title: Promoting Mental and Physical Well-being Through Smart Health
Status: Completed | Type: Observational
Sponsor: IRCCS Centro Neurolesi Bonino Pulejo (Other)
Responsible Party: Principal Investigator, Silvia Marino, Neurologist, IRCCS Centro Neurolesi Bonino Pulejo
Other Study IDs: BRAINHEART22
Record Dates: First submitted 2023-03-13; First posted 2023-03-27 (Actual); Last update posted 2023-03-27 (Actual); Status verified 2023-03

CONDITIONS: Health Behavior; Healthy Lifestyle
MeSH Terms: conditions — Health Behavior

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group 1: All patients are assessed. The neuropsychologist assessed global cognitive status and disposition to Mindfulness. Engineered bands for multi-parameter heart rate monitoring were delivered.From the time of delivery, for 9 consecutive days the patient received a reminder via WhatsApp at the most convenient time slot. At this point, he would wear the supplied chest strap by wetting it appropriately so that it adhered perfectly to the skin. The heart rate App was accessed via Bluetooth and recorded the basal heart rate for about 10 minutes.Then the Mindfulness session was carried out. At the end of 9 days, the completed input tests plus the heart rate measurement were sent on day 10, except for the Mindfulness session, which was not scheduled. After two weeks, the measurement was repeated with the same procedure.
  Interventions: Behavioral: ACT MINDFULNESS
- Group 2: Patients in this group met the inclusion criteria and did not take any measurements. They underwent only the neuropsychological evaluation
  Interventions: Behavioral: ACT MINDFULNESS

INTERVENTIONS:
Behavioral: ACT MINDFULNESS — Mindfulness (MCBT) practices were offered to patients with the aim of fostering the elderly's pro-active role in health prevention by making them
  aware of the relationship between thoughts, emotions and symptomatology of the disorder. The exercises will also be used as a motivational work tool within a protocol of Acceptance and Commitment Therapy (ACT), a new generation cognitive behavioral approach, in which "commitment" components are added to mindfulness, suitable for lifestyle modification.

SUMMARY:
The objective of the study is to develop a smartphone application dedicated to health prevention in terms of monitoring physical activity and healthy eating, mediated by the use of Mindfulness-ACT exercises to reduce unhealthy lifestyles and monitoring through the use of engineered wearable bands.

This is a nonpharmacological prospective observational study. The procedure includes consecutive enrollment in the study of 40 subjects who meet all inclusion criteria. Patients will undergo comprehensive cognitive assessment with collection of all medical history data and information on current clinical condition, including dietary lifestyle. After that they will be invited to register on Brainhearth platform, and then via the app monitoring of physical activity and nutrition, mediated by the use of Mindfulness-ACT exercises, will take place.

DETAILED DESCRIPTION:
The Brainheart study aims to develop a smartphone application connected to a smartwatch dedicated to the prevention of cardiovascular disease among the elderly in their activities of daily living. In addition, to promote health by monitoring physical activity through special engineered bands and healthy eating, mediated by the use of Mindfulness-ACT exercises and appropriate dietary regimen, according to the attached scheme (Appendix A);to acquire physiological and behavioral correlates through the BRAINHEART platform;to develop physical activity, nutrition and interactive exercise programs based on MCBT and ACT; administering contextualized MCBT and ACT cognitive behavioral exercises to promote program adherence;enhancing meta-cognitive skills through a better understanding of the individual with respect to his or her own cognitive processes and their functioning;improving quality of life and one's mental and physical well-being;increasing scientific and clinical knowledge for mental and physical well-being and strategies to promote it;increasing sense of self-efficacy and self-esteem. To achieve these goals, the application developed on a mobile platform, will be designed by integrating:

* a multi-sensory wearable device capable of acquiring and processing physiological and behavioral data to monitor physical and mental health status
* advanced artificial intelligence-based decision support models that can recognize physical and mental health status and provide personalized physical activity and nutrition programs
* exercises and interactive games based on the cognitive behavioral technique Mindfulness and ACT, contextualized and customized in order to increase awareness of health status and motivate the elderly to pursue a healthy lifestyle and best follow the cerebrocardiovascular disease prevention program

STUDY DESIGN.

This is a nonpharmacological prospective observational study.

DURATION OF THE STUDY

Overall, the study will have a duration of 12 months.

STUDY POPULATION

A total of 40 subjects will be consecutively enrolled in the study who are afferent to the facility's outpatient clinics and meet all inclusion criteria, and who will be evaluated at the time of recruitment (T0), and at 6 (T1) and 12 months (T2) intervals. All patients will be assessed by the (a) MMSE, (b) batteries provided within the Brief Neuropsychological Examination, (c) quality of life assessment questionnaires, and (d) Mini Nutritional Assessment (see Annex A to this protocol).

Inclusion criteria

* Age of subjects: 50-85 years.
* Subjects with global cognitive functioning at normal limits (MMSE ≥ 20)
* Subjects with a diagnosis of mild and/or absent depression

Exclusion criteria.

* Diagnosis of dementia
* Diagnosis of moderate/severe depression
* Speech disorders;
* Psychiatric disorders;
* Praxic deficits.

Materials

The project involves the use of:

* portable devices with adequate computational and memory capabilities;
* wireless wearable sensors capable of simultaneously measuring heart rate (HR), and physical activity using triaxial accelerometer;
* mobile processing units for extraction of biosignal features and automatic classification of stress levels.

ELIGIBILITY:
Inclusion Criteria:

- Age of subjects: 50-85 years

* Subjects with global cognitive functioning at normal limits (mmse ≥ 20)
* Subjects with diagnosed mild and/or absent depression;

Exclusion Criteria:

* Diagnosis of dementia
* Diagnosis of moderate/severe depression
* Language disorders
* Psychiatric disorders
* Praxic deficits.

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Forty subjects (20 adult subjects for the experimental group and 20 adult subjects for the control group) were recruited from the Bonino-Pulejo Neurolesi Center in Messina, Italy.
Sampling Method: Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2022-07-27 (Actual); Primary Completion 2022-12-27 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Mindfulness Awareness Attention Scale MAAS | 15 DAYS
  The Mindfulness Awareness Attention Scale measures an individual's tendency for mindfulness in an intentional way, based on the frequency in which he or she is mind-ful or mind-less in his or her experiences.

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Centro Neurolesi "Bonino-Pulejo", Messina, Italy

IPD SHARING:
Plan to Share IPD: No
Corresponding author